CLINICAL TRIAL: NCT07157423
Title: Safety of Eptacog Alfa in Severe Postpartum Haemorrhage in India: A Phase IV Interventional Study
Brief Title: A Research Study to See How Safe is Eptacog Alfa When Used to Stop Heavy Bleeding in Women After Giving Birth in India
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7711-7717; U1111-1289-2568 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-08-19; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Severe Postpartum Haemorrhage
MeSH Terms: conditions — Postpartum Hemorrhage | interventions — recombinant FVIIa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eptacog alfa (NovoSeven) (Experimental): Participants will receive single dose of intravenous bolus injection of eptacog alfa (NovoSeven)
  Interventions: Drug: Eptacog alfa (NovoSeven)

INTERVENTIONS:
Drug: Eptacog alfa (NovoSeven) — Participants will receive single dose of intravenous bolus injection of eptacog alfa (NovoSeven)

SUMMARY:
This study will look at how safe is the medicine eptacog alfa when used in women in India for stopping heavy bleeding after giving birth. If participants have heavy bleeding after giving birth then they will get the medicine eptacog alfa. This study will be conducted to get more knowledge on the safety of the medicine eptacog alfa use in these women. At first participants will receive one dose of medicine eptacog alfa. If the given dose is not helpful to stop the bleeding, participants will get one additional dose. The study will last for about 30-35 days.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study except for blood loss estimation post-partum
* Adult women aged greater than or equal to (≥) 18 years at the time of signing the informed consent and who deliver after 27 weeks diagnosed with severe postpartum haemorrhage (PPH) who fail to respond to uterotonics

Exclusion Criteria:

* Previous participation in this study. Participation is defined as having given informed consent in this study
* Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
* Patient with a history of thromboembolism
* Patient with a history of bleeding disorders
* Patient with a history of or ongoing disseminated intravascular coagulation (DIC); haemolysis, elevated liver enzymes, low platelet count (HELLP) syndrome, thrombotic thrombocytopenic purpura (TTP), pre-eclampsia or other severe complication of childbirth apart from severe PPH
* Have undergone invasive obstetric procedures for the ongoing haemorrhage prior to trial enrolment (uterine balloon tamponade and external aortic compression not included)
* Any chronic disorder or severe disease which, in the opinion of the Investigator, might jeopardise patient's safety or compliance with the protocol
* Participation (i.e., signed informed consent) in any other interventional clinical study prior to screening in the current study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-08-26 (Actual); Primary Completion 2027-03-26 (Estimated); Study Completion 2027-03-26 (Estimated)

PRIMARY OUTCOMES:
Number of thromboembolic events | From baseline (day 0) to end of study (day 30)
  Measured as number of events

SECONDARY OUTCOMES:
Number of serious adverse events | From baseline (day 0) to end of study (day 30)
  Measured as number of events
Number of allergic reactions | From baseline (day 0) to end of study (day 30)
  Measured as number of allergic reactions
All medication errors | Baseline (day 0)
  Measured as number of all medication errors
Near medication errors | Baseline (day 0)
  Measured as number of near medication errors

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (7):
- India (7):
  - KLE Belgum, Belagavi, Karnataka
  - Calicut Medical College, Kozhikode, Kerala
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharashtra
  - SMS Hospital, Jaipur, Rajasthan
  - KLE Belgum, Belagavi
  - Post Graduate Institute of Medical Education & Research_Chandigarh, Chandigarh
  - All India Institute of Medical Sciences_New Dehli, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com